CLINICAL TRIAL: NCT05918120
Title: Screening Using Portable Electronic Recorders for Sleep Apnea in Hypertensive At-Risk Populations (SUPER-SHARP Trial)
Acronym: SUPER-SHARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5749
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: Home Sleep Apnea Tests
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Sleep Apnea Test (Experimental): Patients will undergo assessment for obstructive sleep apnea using a home sleep apnea test.
  Interventions: Device: Home Sleep Apnea Test
- In-laboratory Polysomnography (Active Comparator): Patients receive standard of care for diagnosing obstructive sleep apnea, which is in-laboratory polysomnography.
  Interventions: Device: In-laboratory polysomnography

INTERVENTIONS:
Device: Home Sleep Apnea Test — Use of a home sleep apnea test that records respiratory effort, pulse, oxygen saturation and nasal flow, and reports apneas, hypopneas, flow limitation, snoring and blood oxygen saturation in order to detect obstructive sleep apnea.
  Other Names: HSAT
  Arms: Home Sleep Apnea Test
Device: In-laboratory polysomnography — Level 1 in-laboratory polysomnography for the detection of obstructive sleep apnea.
  Other Names: iPSG
  Arms: In-laboratory Polysomnography

SUMMARY:
Uncontrolled hypertension is associated with an increased risk of heart disease, stroke, and mortality. Obstructive sleep apnea (OSA) is common in hypertension and treatment using continuous positive airway pressure (CPAP) has been shown to effectively lower blood pressure. Despite its clinical significance, OSA remains underdiagnosed in patients with hypertension, because the current standard of care to diagnose OSA is in-laboratory polysomnography, which is inconvenient and often inaccessible for high-risk populations. An alternative to in-laboratory polysomnography is home sleep apnea testing, which has been validated against in-laboratory polysomnography and may be more convenient, accessible, and potentially cost-effective. The objective of this study is to compare home sleep apnea testing to in-laboratory polysomnography in a randomized controlled trial. The investigators will assess whether the use of home sleep apnea testing, compared to use of in-laboratory polysomnography, leads to higher rates of OSA diagnosis and treatment using CPAP, a reduction in blood pressure, improved sleep-related outcomes, and greater patient satisfaction among patients with hypertension at 6 months. The investigators will also assess whether home testing is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* (1) Hypertension, defined as:
* uncontrolled blood pressure on or off medications, or
* controlled blood pressure on 2 or more blood-pressure lowering medications
* (2) At high risk for OSA:
* STOP-BANG sleep apnea screening tool ≥3, or
* Concomitant renal disease (estimated glomerular filtration rate [eGFR] 15-59), or
* Resistant hypertension, defined as a blood pressure above target despite 3 or more BP-lowering drugs at optimal doses (preferably including a diuretic)

Exclusion Criteria:

* prior diagnosis of OSA, current use of CPAP, life expectancy less than 6 months, eGFR<15, gestational hypertension or preeclampsia, current use of dialysis, and physical/cognitive impairment/language barrier restricting the ability to complete the study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of OSA | 6 months
  The investigators will track the number of subjects in each arm who are diagnosed with OSA. Subjects who withdraw or are lost to follow-up without receiving a diagnosis of OSA will be included in our analysis as not having received an OSA diagnosis.

SECONDARY OUTCOMES:
Treatment using CPAP | 6 months
  The proportion of patients treated for OSA using CPAP
Change in 24-hour ambulatory blood pressure | 6 months
  Change in 24-hour ambulatory blood pressure from baseline to 6 months
Sleep-related quality of life (as assessed by the Functional Outcomes of Sleep Questionnaire) | 6 months
  Sleep-related quality of life (as assessed by the Functional Outcomes of Sleep Questionnaire) at 6 months. Functional Outcomes of Sleep Questionnaire (FOSQ) encompasses 5 subscales: activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome. An average score is calculated for each subscale and the 5 subscales are totaled to produce a total score. Subscale scores range from 1-4 with total scores ranging from 5-20. Higher scores indicate better functional status.
Daytime Sleepiness (as assessed by the Epworth Sleepiness Scale) | 6 months
  Daytime Sleepiness (as assessed by the Epworth Sleepiness Scale) at 6 months. Scores on Epworth Sleepiness Scale range from range from 0 to 24, with higher scores indicating higher average sleep propensity in daily life (daytime sleepiness).
Patient satisfaction with sleep testing | 6 months
  Patient satisfaction for each strategy and treatment (as assessed by a Likert scale) at 6 months. Scores range from 0-16, with higher scores indicating increased satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mark I Boulos, MD, MSc, Principal Investigator — University of Toronto and Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Citrus Medical Clinic, Toronto, Ontario